CLINICAL TRIAL: NCT07290478
Title: A Randomized Trial to Encourage Older Adults and Adults With Serious Illness to Designate a Health Care Proxy
Brief Title: Encouraging Older Adults and Adults With Serious Illness to Designate a Health Care Proxy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Contra Costa Health (Unknown)
Responsible Party: Principal Investigator, Mireille Jacobson, Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: UP-23-01203; P30AG024968 (NIH)
Record Dates: First submitted 2025-12-12; First posted 2025-12-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Designating a Healthcare Proxy
Keywords: healthcare proxy; advance care planning; end-of-life care; surrogate decision-maker; durable power of attorney; behavioral economics; pre-commitment

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial + a no intervention control group
Masking Description: Hospital staff, including clinicians, will not be alerted to the patient's assigned intervention. However, clinicians may learn of the patient's assigned intervention if the patient brings their mailer to the visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Personalized Provider Mailer with a Pre-commitment Prompt (Experimental): Patients will receive a mailer containing a pre-commitment prompt to bring in a form listing their healthcare proxy to their next primary care visit. The mailer will be sent from and signed by their primary care provider.
  Interventions: Behavioral: Mailer; Behavioral: Personalized Provider Request; Behavioral: Pre-commitment Prompt
- Generic Health System Mailer with a Pre-commitment Prompt (Experimental): Patients will receive a mailer containing a pre-commitment prompt to bring in a form listing their healthcare proxy to their next primary care visit. The mailer will be sent from and signed by the health system
  Interventions: Behavioral: Mailer; Behavioral: Pre-commitment Prompt
- Personalized Provider Mailer without a Pre-commitment Prompt (Experimental): Patients will receive a mailer, but it will not contain a pre-commitment prompt to bring in a form listing their healthcare proxy to their next primary care visit. The mailer will be sent from and signed by the patient's provider.
  Interventions: Behavioral: Mailer; Behavioral: Personalized Provider Request
- Generic Health System Mailer without a Pre-commitment Prompt (Experimental): Patients will receive a mailer, but it will not contain a pre-commitment prompt to bring in a form listing their healthcare proxy to their next primary care visit. The mailer will be sent from and signed by the health system.
  Interventions: Behavioral: Mailer
- No Mailer Control (No Intervention): Patients will not receive a mailer.

INTERVENTIONS:
Behavioral: Mailer — Patient mailers will ask the patient to name a healthcare proxy at their next primary care visit.
  Arms: Generic Health System Mailer with a Pre-commitment Prompt; Generic Health System Mailer without a Pre-commitment Prompt; Personalized Provider Mailer with a Pre-commitment Prompt; Personalized Provider Mailer without a Pre-commitment Prompt
Behavioral: Personalized Provider Request — Patient mailers will be sent from and signed by the patient's provider for their next scheduled primary care visit.
  Arms: Personalized Provider Mailer with a Pre-commitment Prompt; Personalized Provider Mailer without a Pre-commitment Prompt
Behavioral: Pre-commitment Prompt — Patient mailers will contain a box that asks the patient to bring a form with their choice for a healthcare proxy to their next primary care visit.
  Arms: Generic Health System Mailer with a Pre-commitment Prompt; Personalized Provider Mailer with a Pre-commitment Prompt

SUMMARY:
This study is a Stage III randomized trial to encourage patients in advance of a health care appointment to designate a healthcare proxy. Patients will be randomly assigned to receive a mailer containing information about designating a healthcare proxy, or to not receive any mailer. For patients assigned to receive a mailer, the mailer will differ by the presence or absence of a patient pre-commitment prompt, and contain a personalized provider request or a generic health system request. The work will evaluate the randomized trial and identify factors that predict intervention effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* No EHR-documented healthcare proxy at enrollment
* Age ≥ 55 years OR age ≥ 18 years and listed in the health system's cancer, CHF, or CKD registries

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with EHR-documented healthcare proxy | Within 30 days of the patient's first scheduled primary care visit
  Documentation in the electronic health record of a healthcare proxy

SECONDARY OUTCOMES:
Proportion of patients with EHR-documented advance care planning conversation | Within 30 days of the patient's first scheduled primary care visit
  Documentation in the electronic health record of any advance care planning conversation
Proportion of patients that attended scheduled visit | On the date of the patient's first scheduled primary care visit
  Patient attended the scheduled primary care visit
Proportion of patients with EHR-documented healthcare proxy within 90 days | Within 90 days of the patient's first scheduled primary care visit
  Documentation in the electronic health record of a healthcare proxy
Proportion of patients with EHR-documented advance care planning conversation within 90 days | Within 90 days of the patient's first scheduled primary care visit
  Documentation in the electronic health record of any advance care planning conversation
Proportion of patients with primary care visit within 90 days | Within 90 days of the patient's first scheduled primary care visit
  Patient attended a primary care visit

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Jacobson, PhD, Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD used for results publication may be shared upon request and with approval by the health system.
Supporting Information: SAP, Analytic Code
Time Frame: IPD will be available for one year after the study publication date.
Access Criteria: IPD access criteria will be governed by a data use agreement signed by both parties.